CLINICAL TRIAL: NCT01171339
Title: Prioritising and Optimising Multiple Medications in Elderly Multimorbid Patients in General Practice. - A Pragmatic Cluster-randomised Controlled Trial.
Brief Title: Prioritising and Optimising Multi-medication in Multimorbidity
Acronym: PRIMUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Johann Wolfgang Goethe University Hospital (Other); University Hospital Heidelberg (Other); Heidelberg University (Other); Maastricht University Medical Center (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Christiane Muth, Dr. Chrstiane Muth, MD, MPH, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Muth
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Chronic Disease
Keywords: elderly; multimorbidity; polypharmacy; multimedication; medication appropriateness; medication appropriateness index; cluster-randomised controlled trial; pragmatic trial
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Usual care in accordance with recommended standard#
  #Recommended standard: clinical practice guideline "Geriatrie" of the guideline group of Hesse (part 1 and 2)
- Intervention arm (Experimental): Intervention: Healthcare assistant (HCA) and computer assisted optimization of multi-medication (complex intervention) in accordance with recommended standard#
  #Recommended standard: clinical practice guideline "Geriatrie" of the guideline group of Hesse (part 1 and 2)
  Interventions: Other: Optimization strategy (complex intervention)

INTERVENTIONS:
Other: Optimization strategy (complex intervention) — Healthcare assistant (HCA) and computer assisted optimization of multi-medication (complex intervention) in accordance with recommended standard#
  #Recommended standard: clinical practice guideline "Geriatrie" of the guideline group of Hesse (part 1 and 2)
  Other Names: Intervention arm
  Arms: Intervention arm

SUMMARY:
Objective: To investigate whether the complex intervention will improve the appropriateness of prescriptions in elderly multi-morbid patients with multi-medication in general practices.

Study hypothesis: The primary objective of the study is to determine whether the complex intervention will improve the appropriateness of prescriptions compared to usual care. The primary efficacy endpoint is the change in the Medication Appropriateness Index (MAI) score from baseline (T0) to 6 months after baseline (T1), i.e. the difference MAI T1-T0.

DETAILED DESCRIPTION:
Key elements (1 to 4) of the complex intervention:

1. Basic assessment of medicines that were actually taken (brown bag review) by a general practice based health care assistant (HCA) and
2. Checklist-based (MediMoL - Medication-Monitoring-List) pre-consultation interview on problems relating to medicines (technical handling, potential adverse drug reactions) and patient's therapeutic aims by HCA provides structured information in the Medication-Monitoring-List (MediMoL) for the general practitioner (GP) and enables patients to discuss their problems with the GP.
3. GP uses a computerized decision support system (pharmaceutical information system, AiD+) to optimize medication (reducing number of inappropriate prescriptions, e.g. pharmaceutical interactions, renal dose adjustments, duplicate prescriptions) and
4. prioritizes medication in the physician-patient consultation taking into consideration patient's preferences.

ELIGIBILITY:
Inclusion Criteria:

* at least 60 years old of both sexes
* at least three chronic diseases affecting two or more organ systems, which require pharmaceutical treatment
* at least five long-term prescriptions with systemic effects
* health care provided by GP (at least one contact in most recent quarter)
* patient is legally competent to sign any documents
* ability to understand and participate in trial of own free will, to fill out questionnaires and participate in telephone interviews
* written informed consent to participate in trial

Exclusion Criteria:

* diseases cause life expectancy of less than 12 months
* abuse of alcohol or illegal drugs and visible clinical signs or symptoms thereof
* cognitive impairment that prevents trial participation (MMSE < 26)
* emotional stress that prevents trial participation
* participation in a clinical trial within the last 30 days

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-02-29 (Actual)

PRIMARY OUTCOMES:
Medication Appropriateness Index (MAI)-Score | 6 months from baseline
  Difference in Medication Appropriateness Index (MAI)-Score 6 months from baseline minus baseline (MAI T1-T0)

SECONDARY OUTCOMES:
MAI-Score | 9 months from baseline
  Difference in Medication Appropriateness Index (MAI)-Score 9 months from baseline minus baseline (MAI T1-T0)
Generic health related quality of life: EQ-5D | 6 months from baseline
  Change in generic health related quality of life measured as the difference in the EQ-5D-Score 6 months from baseline minus baseline (T1-T0)
Generic health related quality of life: EQ-5D | 9 months
  Change in generic health related quality of life measured as the difference in the EQ-5D-Score 9 months from baseline minus baseline (T2-T0)
Functional disability: Vulnerable Elderly Survey (VES-13) | 6 months
  Change in functional disability measured as the difference in the VES-13-Score 6 months from baseline minus baseline (T1-T0)
Functional disability: Vulnerable Elderly Survey (VES-13) | 9 months
  Change in functional disability measured as the difference in the VES-13-Score 9 months from baseline minus baseline (T2-T0)
Change in all cause hospitalisation | 6 months and 9 months
"Observed" adherence | 6 months from baseline and 9 months from baseline
  Change in observed adherence measured as the difference between intake (patient's interview) and prescribed medication (CRF reported by physician's) 6 months from baseline minus baseline (T1-T0) and 9 months from baseline minus baseline (T2-T0)
Self-reported adherence (Morisky) | 6 and 9 months from baseline
  Change in self-reported adherence measured as the difference in the Morisky-Score 6 months from baseline minus baseline (T1-T0) and 9 months from baseline minus baseline (T2-T0)
Future life expectancy / years of desired life | 6 and 9 months from baseline
  Change in perceived future life expectancy reflects concepts of will to life or years of desired life [YDL] measured as the difference of the three items future expectation / expected lifetime duration / desired lifetime duration in the interval 6 months
medication complexity | 6 and 9 months from baseline
  Change in complexity of medication measured as the difference 6 months from baseline minus baseline (T1-T0) and 9 months from baseline minus baseline (T2-T0)
  * Total number of prescriptions
  * Number of single doses / day
  * Medication Regimen Complexity Index (MRCI)
Beliefs about Medicines Questionaire (BMQ) | 6 and 9 months from baseline
  Change in health and illness beliefs and attitudes measured as the difference in the Beliefs about Medicines Questionaire (BMQ) score 6 months from baseline minus baseline (T1-T0) and 9 months from baseline minus baseline (T2-T0)
Severity of chronic pain | 6 and 9 months from baseline
  Change in severity of chronic pain measured as the difference in Characteristic Pain Intensity score, the Disability Score, in Disability Points and the resulting Grades of chronic pain severity in accordance with M. von Korff, J. Ormel et al. the interval 6 months from baseline minus baseline (T1-T0) and 9 months from baseline minus baseline (T2-T0)
Satisfaction with shared decision making (Man Son Hing scale, MSH) | 6 and 9 months from baseline
  Change in satisfaction with shared decision making measured as the difference in the Man Son Hing scale (MSH) interval 6 months from baseline minus baseline (T1-T0) and 9 months from baseline minus baseline (T2-T0)
Cognitive dysfunction in verbal fluency | 6 and 9 months from baseline
  Change in cognitive (dys)function measured as the difference in the Verbal Fluency Test (VFT) interval 6 months from baseline minus baseline (T1-T0) and 9 months from baseline minus baseline (T2-T0)
Depressive symptoms | 6 and 9 months from baseline
  Change in depressive symptoms measured as the difference in the Geriatric Depression Scale (GDS) interval 6 months from baseline minus baseline (T1-T0) and 9 months from baseline minus baseline (T2-T0)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Muth, MD, MPH, Principal Investigator — Institute for General Practice, Goethe-University Frankfurt / Main
Locations (1):
- Institute for General Practice, Goethe-University Frankfurt / Main, Germany, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Buedingen F, Hammer MS, Meid AD, Muller WE, Gerlach FM, Muth C. Changes in prescribed medicines in older patients with multimorbidity and polypharmacy in general practice. BMC Fam Pract. 2018 Jul 28;19(1):131. doi: 10.1186/s12875-018-0825-3. PMID 30055583
- [Derived] Muth C, Uhlmann L, Haefeli WE, Rochon J, van den Akker M, Perera R, Guthlin C, Beyer M, Oswald F, Valderas JM, Knottnerus JA, Gerlach FM, Harder S. Effectiveness of a complex intervention on Prioritising Multimedication in Multimorbidity (PRIMUM) in primary care: results of a pragmatic cluster randomised controlled trial. BMJ Open. 2018 Feb 24;8(2):e017740. doi: 10.1136/bmjopen-2017-017740. PMID 29478012